CLINICAL TRIAL: NCT07004569
Title: A Prospective, Non-Randomized, Clinical Registry of The AngioliteTM Durable Fluoroacrylate Polymer-based Sirolimus-Eluting Stent in The Treatment of Patients With Left Main Coronary Artery Lesions
Brief Title: Angiolite Registry Study
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2024.682
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: With Left Main Coronary Artery Lesions
Keywords: Polymer-based Sirolimus-Eluting Stent
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using AngioliteTM Stent with Left Main Coronary Artery Lesions: This is an investigator-initiated, prospective, single-centre, non-randomized registry that evaluates the safety and efficacy of the AngioliteTM Durable Fluoroacrylate Polymer-based Sirolimus-Eluting Stent (iVascular, Barcelona, Spain) for the treatment of LMCA disease.
  Interventions: Device: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — Patients is under Percutaneous coronary intervention (PCI) by using contemporary drug eluting stent (DES). Angiolite is a thin-strut cobalt-chromium durable fluoroacrylate polymer-based, sirolimus-eluting stent that is CE marked and commercially available. Stent sizes 2.0mm to 4.5mm in 9mm to 49mm lengths will be used.

SUMMARY:
Left main coronary artery (LMCA) is a major branch of coronary artery and supplies a large bulk of myocardium. Percutaneous coronary intervention (PCI) using contemporary drug eluting stent (DES) is one of the treatment options for patients with significant LMCA disease and suitable anatomy as multiple randomized controlled trials and meta-analysis have demonstrated the feasibility and safety of PCI in the treatment of LMCA disease. There are a few challenges in LMCA PCI due to certain anatomical and structural factors. The LMCA disease frequently involves bifurcations which requires special considerations such as side-branch access and preservation in order to prevent procedural related myocardial infarction (MI). Implantation of a metallic scaffold across the LMCA bifurcation often requires aggressive post-dilatation of the LMCA stent due to the diameter discrepancy between the side-branch and the LMCA main body. However, overexpansion beyond the rated diameter might compromise the stent integrity and radial force, resulting in mal-apposition, vascular recoil and risk of subsequent target lesion failure (TLF). The Angiolite stent is a thin-strut cobalt-chromium sirolimus-eluting stent with an open-cell design and a high overexpansion capacity that might overcomes some of these challenges in LMCA PCI. The ANGIOLITE randomized trial confirmed the non-inferiority of the Angiolite stent against the conventional DES. However, patients with LMCA involvement were specifically excluded from the trial. We therefore propose to investigate the procedural and 24 months clinical performance of the Angiolite stent in the treatment of patients with LMCA lesions.

DETAILED DESCRIPTION:
Left main coronary artery (LMCA) is a major branch of coronary artery and supplies a large bulk of myocardium. Percutaneous coronary intervention (PCI) using contemporary drug eluting stent (DES) is one of the treatment options for patients with significant LMCA disease and suitable anatomy as multiple randomized controlled trials and meta-analysis have demonstrated the feasibility and safety of PCI in the treatment of LMCA disease. There are a few challenges in LMCA PCI due to certain anatomical and structural factors. The LMCA disease frequently involves bifurcations which requires special considerations such as side-branch access and preservation in order to prevent procedural related myocardial infarction (MI). Implantation of a metallic scaffold across the LMCA bifurcation often requires aggressive post-dilatation of the LMCA stent due to the diameter discrepancy between the side-branch and the LMCA main body. However, overexpansion beyond the rated diameter might compromise the stent integrity and radial force, resulting in mal-apposition, vascular recoil and risk of subsequent target lesion failure (TLF). The Angiolite stent is a thin-strut cobalt-chromium sirolimus-eluting stent with an open-cell design and a high overexpansion capacity that might overcomes some of these challenges in LMCA PCI. The ANGIOLITE randomized trial confirmed the non-inferiority of the Angiolite stent against the conventional DES. However, patients with LMCA involvement were specifically excluded from the trial. We therefore propose to investigate the procedural and 24 months clinical performance of the Angiolite stent in the treatment of patients with LMCA lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age >18.
2. Subject (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent.
3. Indication for a percutaneous coronary intervention (PCI) in native epicardial arteries involving left main coronary artery, including patients with stable coronary artery disease and acute coronary syndromes (non-ST-elevated myocardial infarction and ST-elevation myocardial infarction).
4. Target lesion must have a stenosis of >50% and <100% angiographically.
5. Target lesion much have an angiographic reference vessel diameter of 2.0-6.0 mm.
6. All lesions requiring PCI should be amendable for implantation of study stents.

Exclusion Criteria:

1. Known history of an allergic reaction or significant sensitivity to sirolimus or other analogue or derivative.
2. Known history of an allergic reaction or significant sensitivity to fluoroacrylate or its analogue or derivative.
3. Pregnant or breastfeeding woman.
4. Currently participating in another device study that has not completed the primary end point or that clinically interferes with the current study endpoints.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include up to 50 patients of both genders who meet the eligibility criteria listed below and agree to participate in the trial
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
change in Device oriented clinical endpoint (DOCE) | baseline, 1 month, 6 months, 12 months, 24 months
  Device oriented clinical endpoint (DOCE) defined as a composite of cardiovascular death, myocardial infarction (Q-wave and non-Q wave), emergent coronary artery bypass graft surgery, target vessel myocardial infarction (TV-MI) or repeat clinically driven target-lesion revascularization (TLR) by percutaneous or surgical methods.

OTHER OUTCOMES:
Lesion successful rate | baseline, 1 month, 6 months, 12 months, 24 months
  Lesion successful rate is achieving less than 30% residual stenosis on angiography after the usage of the study device with lesion preparation and post-dilatation.
Device successful rate | baseline, 1 month, 6 months, 12 months, 24 months
  Device successful rate is successful implantation of the study device at the target lesions
Procedural successful rate | baseline, 1 month, 6 months, 12 months, 24 months
  Procedural successful rate is lesion success and no DOCE during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong